CLINICAL TRIAL: NCT02241161
Title: Short Term Evaluation of the Soothing and Re-epithelizing Activity of Three Topical Products and Relative Combinations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2913
Record Dates: First submitted 2014-07-18; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: skin eythema; rejuvenating cream; rejuvenating serum; antioxidant serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- plantaricin a - rejuvenating cream (Active Comparator): single application on an area of 17,5 cm2, on the forearm, after skin stripping, and left absorbing on the skin for at least 15 minutes
  Interventions: Other: plantaricin a - rejuvenating cream
- plantaricin a - rejuvenating serum (Active Comparator): single application on an area of 17,5 cm2, on the forearm, after skin stripping, and left absorbing on the skin for at least 15 minutes
  Interventions: Other: plantaricin a - rejuvenating serum
- plantaricin a - antioxidant serum (Active Comparator): single application on an area of 17,5 cm2, on the forearm, after skin stripping, and left absorbing on the skin for at least 15 minutes
  Interventions: Other: plantaricin a - antioxidant serum
- plantaricin a (rejuvenating cream +rejuvenating serum) (Active Comparator): single application on an area of 17,5 cm2, on the forearm, after skin stripping, and left absorbing on the skin for at least 15 minutes
  Interventions: Other: plantaricin a - rejuvenating cream; Other: plantaricin a - rejuvenating serum
- plantaricin a (rejuvenating cream + antioxidant serum) (Active Comparator): single application on an area of 17,5 cm2, on the forearm, after skin stripping, and left absorbing on the skin for at least 15 minutes
  Interventions: Other: plantaricin a - rejuvenating cream; Other: plantaricin a - antioxidant serum

INTERVENTIONS:
Other: plantaricin a - rejuvenating cream — single application on an area of 17,5 cm2, on the forearm, after skin stripping, and left absorbing on the skin for at least 15 minutes
  Arms: plantaricin a (rejuvenating cream + antioxidant serum); plantaricin a (rejuvenating cream +rejuvenating serum); plantaricin a - rejuvenating cream
Other: plantaricin a - antioxidant serum — single application on an area of 17,5 cm2, on the forearm, after skin stripping, and left absorbing on the skin for at least 15 minutes
  Arms: plantaricin a (rejuvenating cream + antioxidant serum); plantaricin a - antioxidant serum
Other: plantaricin a - rejuvenating serum — single application on an area of 17,5 cm2, on the forearm, after skin stripping, and left absorbing on the skin for at least 15 minutes
  Arms: plantaricin a (rejuvenating cream +rejuvenating serum); plantaricin a - rejuvenating serum

SUMMARY:
Aim of the study was to evaluate the soothing and re-epithelizing activity of a single application of topical products on experimentally induced erythema by skin stripping on the forearm (volar surface) of 20 healthy volunteers. In particular the activity of the following three cosmetic products and the relative combinations (cream and serum) were assessed: rejuvenating cream, rejuvenating serum, antioxidant serum

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers of both sexes, aged more than 18 years old
* Volunteers in a good general state of health in the Investigator opinion
* Volunteers not taking drugs or undergoing surgical procedure
* Volunteers who are giving a written informed consent.

Exclusion Criteria:

* Pregnancy (only for female subjects)
* lactation (only for female subjects)
* change in the normal habits in the last month
* participation in a similar study during the previous month
* known allergy to one or several ingredients of the products on trial
* insufficient adhesion to the study protocol
* dermatological disease
* clinical and significant skin condition on the test area (e.g. lesions, scars, malformations)
* diabetes
* endocrine disease
* hepatic, renal or cardiac disorder
* cancer
* topical drugs or surgical procedure on the test areas during the previous 3 months
* systemic corticosteroids
* aspirin or non-steroid anti-inflammatory drugs (FANS)
* diuretic drugs
* antibiotics and chemotherapics
* pshycotropic drugs
* retinoids
* psoralens
* cardiologic and vascular drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of skin erythema: change from baseline, 1 hour after products application (T1h vs. T0) | After 1 (T1h) hour from products application
  Skin erythema was scored and recorded according to the following grades: 0=no erythema; 0.5=very slight erythema (barely perceptible);1=well-defined erythema;1.5=moderate to severe erythema; 2=severe erythema (beet redness) to slight eschar formation (injuries in depth)

SECONDARY OUTCOMES:
Clinical evaluation of skin erythema: change from baseline, 6 hours from products application (T6h vs. T0) | After 6 (T6h) hours from products application
  Skin erythema was scored and recorded according to the following grades: 0=no erythema; 0.5=very slight erythema (barely perceptible);1=well-defined erythema;1.5=moderate to severe erythema; 2=severe erythema (beet redness) to slight eschar formation (injuries in depth)
Clinical evaluation of skin erythema: change from baseline, after 24 hours from products application (T24h vs. T0) | After 24 (T24h) hours from products application
  Skin erythema was scored and recorded according to the following grades: 0=no erythema; 0.5=very slight erythema (barely perceptible);1=well-defined erythema;1.5=moderate to severe erythema; 2=severe erythema (beet redness) to slight eschar formation (injuries in depth)
Optical densitometry: change from baseline, after 1hour from products application (T1h vs. T0) | After 1 (T1h) hour from products application
  The instrumental measurement of erythema was performed by the use of an optical densitometer allowing to quantify, on a logarithmic scale, total reflected optical density (visual=V) and the values of primary subtractive colours of reflected light: cyan(=C), magenta(=M) and yellow(=Y). Calculation of erythema index was done as follows: E.I.=logRmagenta-logRcyan
Optical densitometry: change from baseline, 6 hours from products application (T6h vs. T0) | After 6 (T6h) hours from products application
  The instrumental measurement of erythema was performed by the use of an optical densitometer allowing to quantify, on a logarithmic scale, total reflected optical density (visual=V) and the values of primary subtractive colours of reflected light: cyan(=C), magenta(=M) and yellow(=Y). Calculation of erythema index was done as follows: E.I.=logRmagenta-logRcyan
Optical densitometry: change from baseline, 24 hours from products application (T24h vs.T0) | After 24 (T24h) hours from products application
  The instrumental measurement of erythema was performed by the use of an optical densitometer allowing to quantify, on a logarithmic scale, total reflected optical density (visual=V) and the values of primary subtractive colours of reflected light: cyan(=C), magenta(=M) and yellow(=Y). Calculation of erythema index was done as follows: E.I.=logRmagenta-logRcyan
Surface microrelief evaluation: change from baseline, after 1 hour from products application (T1h vs.T0) | After 1 (Th1) hour from products application
  Morfometrical analysis of cutaneous surface allows the evaluation of the regularity of the microrelief (superficial cutaneous network). It was therefore possible to determinate the alteration of the microrelief caused by stripping.The evaluation of the regularity grade of cutaneous microrelief was possible using Fast Fourier Transform (FFT) on skin replicas obtained using silicone rubber. Skin replicas images were then acquired by a stereo microscope.
Surface microrelief evaluation: change from baseline, 6 hours from products application (T6h vs. T0) | After 6 (T6h) hours from products application
  Morfometrical analysis of cutaneous surface allows the evaluation of the regularity of the microrelief (superficial cutaneous network). It was therefore possible to determinate the alteration of the microrelief caused by stripping.The evaluation of the regularity grade of cutaneous microrelief was possible using Fast Fourier Transform (FFT) on skin replicas obtained using silicone rubber. Skin replicas images were then acquired by a stereo microscope.
Surface microrelief evaluation: change from baseline, after 24 hours from products application (T24h) hours from products application vs.T0) | After 24 hours (T24h) from products application
  Morfometrical analysis of cutaneous surface allows the evaluation of the regularity of the microrelief (superficial cutaneous network). It was therefore possible to determinate the alteration of the microrelief caused by stripping.The evaluation of the regularity grade of cutaneous microrelief was possible using Fast Fourier Transform (FFT) on skin replicas obtained using silicone rubber. Skin replicas images were then acquired by a stereo microscope.

CONTACTS AND LOCATIONS:
Overall Officials: Adele Sparavigna, Doctor, Principal Investigator — Derming SRL
Locations (1):
- DermIng SRL, Monza, Monza, Italy

REFERENCES:
- [Background] Buonocore D, Lazzeretti A, Tocabens P, Nobile V, Cestone E, Santin G, Bottone MG, Marzatico F. Resveratrol-procyanidin blend: nutraceutical and antiaging efficacy evaluated in a placebocontrolled, double-blind study. Clin Cosmet Investig Dermatol. 2012;5:159-65. doi: 10.2147/CCID.S36102. Epub 2012 Oct 5. PMID 23071399
- [Background] Benzie IF, Strain JJ. The ferric reducing ability of plasma (FRAP) as a measure of "antioxidant power": the FRAP assay. Anal Biochem. 1996 Jul 15;239(1):70-6. doi: 10.1006/abio.1996.0292. PMID 8660627
- [Background] Bradford MM. A rapid and sensitive method for the quantitation of microgram quantities of protein utilizing the principle of protein-dye binding. Anal Biochem. 1976 May 7;72:248-54. doi: 10.1016/0003-2697(76)90527-3. No abstract available. PMID 942051
- [Background] Calcabrini C, De Bellis R, Mancini U, Cucchiarini L, Potenza L, De Sanctis R, Patrone V, Scesa C, Dacha M. Rhodiola rosea ability to enrich cellular antioxidant defences of cultured human keratinocytes. Arch Dermatol Res. 2010 Apr;302(3):191-200. doi: 10.1007/s00403-009-0985-z. Epub 2009 Aug 25. PMID 19705137
- [Background] Corcuff P, Chatenay F, Leveque JL. A fully automated system to study skin surface patterns. Int J Cosmet Sci. 1984 Aug;6(4):167-76. doi: 10.1111/j.1467-2494.1984.tb00373.x. PMID 19467109
- [Background] De Jongh CM, Verberk MM, Withagen CE, Jacobs JJ, Rustemeyer T, Kezic S. Stratum corneum cytokines and skin irritation response to sodium lauryl sulfate. Contact Dermatitis. 2006 Jun;54(6):325-33. doi: 10.1111/j.0105-1873.2006.00848.x. PMID 16787454
- [Background] Int J Cosm Sci 6: 167-186, 1984 Fernay, Voltaire The World Medical Association (1989)
- [Background] Elsner P, Barel AO, Berardesca E, Gapard B, Serup J Skin Bioengineering Techniques and Applications in Dermatology and Cosmetology Karger, 1998
- [Background] Fuga GC, Spina C, Cavallotti C, Di Palma A, Lombardi G, Marmo W Computerized reflected optical densitometry. A research on the colour of the skin. Journal of Applied Cosmetology, 8:91-110,1990
- [Background] Fullerton A, Fischer T, Lahti A, Wilhelm KP, Takiwaki H, Serup J. Guidelines for measurement of skin colour and erythema. A report from the Standardization Group of the European Society of Contact Dermatitis. Contact Dermatitis. 1996 Jul;35(1):1-10. doi: 10.1111/j.1600-0536.1996.tb02258.x. PMID 8896947
- [Background] Garcia Ortiz P, Hansen SH, Shah VP, Menne T, Benfeldt E. Impact of adult atopic dermatitis on topical drug penetration: assessment by cutaneous microdialysis and tape stripping. Acta Derm Venereol. 2009;89(1):33-8. doi: 10.2340/00015555-0562. PMID 19197539
- [Background] Grove GL, Zerweck CR, Houser TP, Smith GE, Koski NI. A randomized and controlled comparison of gentleness of 2 medical adhesive tapes in healthy human subjects. J Wound Ostomy Continence Nurs. 2013 Jan-Feb;40(1):51-9. doi: 10.1097/WON.0b013e318276f2a4. PMID 23202590
- [Background] ICH Harmonised Tripartite Guideline - Guideline for Good Clinical Practice International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use: May 1996
- [Background] Lademann J, Meinke MC, Schanzer S, Richter H, Darvin ME, Haag SF, Fluhr JW, Weigmann HJ, Sterry W, Patzelt A. In vivo methods for the analysis of the penetration of topically applied substances in and through the skin barrier. Int J Cosmet Sci. 2012 Dec;34(6):551-9. doi: 10.1111/j.1468-2494.2012.00750.x. Epub 2012 Sep 25. PMID 22957937
- [Background] Lademann J, Jacobi U, Surber C, Weigmann HJ, Fluhr JW. The tape stripping procedure--evaluation of some critical parameters. Eur J Pharm Biopharm. 2009 Jun;72(2):317-23. doi: 10.1016/j.ejpb.2008.08.008. Epub 2008 Aug 19. PMID 18775778
- [Background] Lindemann U, Wilken K, Weigmann HJ, Schaefer H, Sterry W, Lademann J. Quantification of the horny layer using tape stripping and microscopic techniques. J Biomed Opt. 2003 Oct;8(4):601-7. doi: 10.1117/1.1609200. PMID 14563197
- [Background] Marttin E, Neelissen-Subnel MT, De Haan FH, Bodde HE. A critical comparison of methods to quantify stratum corneum removed by tape stripping. Skin Pharmacol. 1996;9(1):69-77. doi: 10.1159/000211392. PMID 8868035
- [Background] Sachs L Applied statistics: a handbook of techniques. Heidelberg: Springer, 1981:536-539
- [Background] Serup J, Agner T. Colorimetric quantification of erythema--a comparison of two colorimeters (Lange Micro Color and Minolta Chroma Meter CR-200) with a clinical scoring scheme and laser-Doppler flowmetry. Clin Exp Dermatol. 1990 Jul;15(4):267-72. doi: 10.1111/j.1365-2230.1990.tb02087.x. PMID 2208776
- [Background] Takiwaki H. Measurement of skin color: practical application and theoretical considerations. J Med Invest. 1998 Feb;44(3-4):121-6. PMID 9597799
- [Background] Weigmann H, Lademann J, Meffert H, Schaefer H, Sterry W. Determination of the horny layer profile by tape stripping in combination with optical spectroscopy in the visible range as a prerequisite to quantify percutaneous absorption. Skin Pharmacol Appl Skin Physiol. 1999 Jan-Apr;12(1-2):34-45. doi: 10.1159/000029844. PMID 10325582
- See also: Investigation Center — http://www.derming.com
- See also: Sponsor — http://www.giulianipharma.com/